CLINICAL TRIAL: NCT03726567
Title: Environmental Chemicals That Accumulate in Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/H1304/13
Record Dates: First submitted 2017-07-22; First posted 2018-10-31 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Participants who are undergoing bariatric surgery and control group who is having abdominal surgery for non-bariatric reasons
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bariatric surgery group (Active Comparator): Patients who are undergoing bariatric surgery for weight loss
  Interventions: Procedure: Bariatric surgery
- Non bariatric surgery group (No Intervention): Patients who are undergoing abdominal surgery for non-weight loss reasons

INTERVENTIONS:
Procedure: Bariatric surgery — Roux-en-Y surgery
  Arms: Bariatric surgery group

SUMMARY:
A crucial factor in evaluating the risk of dioxins, and related endocrine disruptor compounds (dioxins for short) in the human population is the accumulation of these chemicals in the human body. Human data on tissue background levels is extremely limited, and there are no studies in UK populations, although there are several European studies looking at blood levels of dioxins. Adipose tissue concentrations were 139 ng of TEQ (total dioxin-like compounds) per kg lipid weight (5.4 ± 4.6 ng of TCDD per kg lipid weight). However, given the different dietary habits of Japanese populations, compared to European populations, these estimates may differ considerably from UK values. Thus determining human tissue concentrations of dioxins is an important issue for assessing the risk to public health from these compounds, and this information is currently lacking for European populations. This information will also guide and inform the necessity fro continued measures to reduce the environmental dioxin levels in the UK.

Aims

Primary outcomes:

1. Investigation of the toxicodynamics of/dioxin distribution in adipose of a morbidly obese and comparative control population
2. Characterisation of the burden of dioxins in liver and adipose tissue, and the relationship with blood levels of dioxins, in a UK population

Secondary outcome:

Determining whether bariatric surgery-induced weight loss causes an increase in tissue concentration of dioxin-like compounds

The primary aims of this study will yield useful information to refine the risk assessment process for the obese population.

Experimental Methodology This proposal seeks to examine thirty non-obese patients taking liver (500mg) and adipose tissue (visceral and subcutaneous: 40g each) samples at the time of gastric/abdominal surgery; and thirty obese patients, taking liver (500mg) and adipose tissue (visceral and subcutaneous: 40g each) samples at the time of undertaking Roux -en-y bariatric surgery. Weight and bioimpedance and a food diary will be performed prior to surgery.

A further body weight and bioimpedance will be undertaken at 3, 6, 9 and 12 months from the obese population. A subcutaneous adipose biopsy will be taken under local anaesthetic from these individuals at after bariatric surgery (minimum of 10% body weight loss). A record of weight loss since bariatric surgery will documented with the change in body composition. The statistical power for seeing an effect of gastroplasty, assuming a coefficient of variation of TEQ measurements of 75% and an increase in TEQ of two-fold, is 90% at P<0.05 for a population of thirty individuals.

Should subjects need additional surgery (eg. cholecystectomy, diagnostic laproscopy) either as a consequence of bariatric surgery or for any other reasons during the 24 month following initial operation, a liver biopsy and visceral fat biopsy will be taken during the future surgery. If subjects undergo abdominal wall surgeries (eg. Apronectomy, ventral hernia repair) in the 24 months following initial bariatric surgery, an subcutaneous fat biopsy will be taken during the future surgery.

DETAILED DESCRIPTION:
Background A crucial factor in evaluating the risk of dioxins, and related endocrine disruptor compounds (dioxins for short) in the human population is the accumulation of these chemicals in the human body. The "half-life" of the prototypical dioxin, 2,3,7,8-tetrachlorodibenzo-p-dioxin (TCDD) in the human is estimated as ~7 years, as such accumulation of these chemicals in the body is an important issue. These lipophilic chemicals accumulate in adipose tissue, and (in a congener-dependent fashion) in the liver, so an accurate estimation of human body burden requires knowledge of their concentrations in liver, and adipose tissue. The concentration of these endocrine disruptors in blood is an essential piece of information for understanding how these chemicals dispose between the organs, and for calibrating tissue concentrations to the most common measurement of dioxins and in humans, which is a measurement of dioxins in blood.

However, human data on tissue background levels is extremely limited, and I am unaware of any studies in UK populations, although there are several European studies looking at blood levels of dioxins. There is one study in an American population, which features some people with a history of (presumably occupational) exposure to TCDD, but this was published in 1988, when background levels were considerably higher. Adipose tissue concentrations were 83 ± 178 ng of TCDD per kg lipid weight. There are three recent studies from Japan, spanning 1999-2007, so these should be indicative of the much lower current background level of dioxin exposure. Adipose tissue concentrations were 139 ng of TEQ (total dioxin-like compounds) per kg lipid weight (5.4 ± 4.6 ng of TCDD per kg lipid weight). However, given the different dietary habits of Japanese populations, compared to European populations, these estimates may differ considerably from UK values. Thus determining human tissue concentrations of dioxins is an important issue for assessing the risk to public health from these compounds, and this information is currently lacking for European populations. This information will also guide and inform the necessity fro continued measures to reduce the environmental dioxin levels in the UK.

A further topical issue relates to the body burden of dioxins in obese individuals, since an increased BMI is associated with increased blood concentration of dioxin and other lipophilic contaminants, and the impact of weight reduction upon the concentration and amount of dioxins in the body is unknown. There is the possibility that weight reduction could result in the release of dioxins from adipose tissue depots, as the adipose tissue is lost, and that the circulating dioxin levels (and other toxic lipophilic chemicals) could increase if the dioxin is maintained in the body, or alternatively as adipose tissue is lost dioxins may be concentrated in the remaining adipose tissue. Although there is some evidence that weight loss is associated with an increase in some lipophilic contaminants, dioxins have not been examined to see if these are increased after weight loss. If dioxin concentrations in lipids increase following weight loss, it will also be useful to evaluate whether those increased concentrations persist or rapidly equilibrate, and the data from this study may allow some evaluation of that question as well. The toxicodynamics information will allow estimation and prediction of what will happen to other lipophilic chemicals in the body.

Aims

Primary outcomes:

1. Investigation of the toxicodynamics of/dioxin distribution in adipose of a morbidly obese and comparative control population
2. Characterisation of the burden of dioxins in liver and adipose tissue, and the relationship with blood levels of dioxins, in a UK population

Secondary outcome:

Determining whether bariatric surgery-induced weight loss causes an increase in tissue concentration of dioxin-like compounds

The primary aims of this study will yield useful information to refine the risk assessment process for the obese population.

Experimental Methodology This proposal seeks to examine thirty non-obese patients taking liver (500mg) and adipose tissue (visceral and subcutaneous: 40g each) samples at the time of gastric/abdominal surgery; and thirty obese patients, taking liver (500mg) and adipose tissue (visceral and subcutaneous: 40g each) samples at the time of undertaking Roux -en-y bariatric surgery. Weight and bioimpedance and a food diary will be performed prior to surgery.

A further body weight and bioimpedance will be undertaken at 3, 6, 9 and 12 months from the obese population. A subcutaneous adipose biopsy will be taken under local anaesthetic from these individuals after bariatric surgery (minimum of 10% body weight loss). A record of weight loss since bariatric surgery will documented with the change in body composition. The statistical power for seeing an effect of gastroplasty, assuming a coefficient of variation of TEQ measurements of 75% and an increase in TEQ of two-fold, is 90% at P<0.05 for a population of thirty individuals.

Should subjects need additional surgery (eg. cholecystectomy, diagnostic laproscopy) either as a consequence of bariatric surgery or for any other reasons during the 24 month following initial operation, a liver biopsy and visceral fat biopsy will be taken during the future surgery. If subjects undergo abdominal wall surgeries (eg. Apronectomy, ventral hernia repair) in the 24 months following initial bariatric surgery, an subcutaneous fat biopsy will be taken during the future surgery.

Measurement of dioxins and TEQ will be performed with high resolution GC-MS in a laboratory accredited for working with dioxins, according to ISO17025. The method is validated to have high sensitivity (necessary for the small volumes of clinical samples) and robust quality control (essential for analyses of background levels of dioxins), and the analytical team have extensive experience of using this technology with demanding biological samples. Lipid content of sampled tissues will also be measured to allow assessment of lipid-adjusted tissue concentrations for comparison across tissues and blood, as previous work has demonstrated that these compounds partition across tissues principally on the basis of lipid content.

Statistical analysis of the effect of gastroplasty on dioxin burden and concentrations will use a conventional repeated measures methodology. Modelling the relationship between tissue distribution and blood concentrations of dioxins, especially with regard to different congeners, will be undertaken by Summit Toxicology, who have extensive experience of these analyses. The data will be evaluated in the framework of a previously-published toxicokinetic model, and potential congener-specific differences in behaviour will be evaluated.

It is anticipated that initial data analysis will be undertaken comparing the dioxin burden between the obese and non-obese subjects (per gram tissue on a wet weight and on a lipid-adjusted basis, and related to lean body mass). The final data analysis will also take into account the change in dioxins with time associated with loss of body weight/change in lean body mass, together with the dioxin load in subcutaneous fat tissue before and after weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of more than 25
* Listed for bariatric surgery
* Control group - participants who are listed for abdominal surgery for non-weight loss reason

Exclusion Criteria:

* Participants unable to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-10-12 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2016-01-30 (Actual)

PRIMARY OUTCOMES:
Concentration of the dioxin and related compounds (endocrine disrupting chemicals) in adipose tissue and liver samples of obese population compared to non-obese population | 2 years
  to investigate the distribution of endocrine disrupting chemicals in obese and control population

SECONDARY OUTCOMES:
Endocrine disrupting chemical concentrations in adipose tissue and liver samples after bariatric surgery | 2 years
  endocrine disrupting chemical concentrations will be measured before and after bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thozhukat Sathyapalan, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Hull and east Yorkshire Hospitals NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Will be published in Food Standards Agency website